CLINICAL TRIAL: NCT00176254
Title: Paclitaxel, Carboplatin and Radiotherapy as Induction Therapy in Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Susanne Arnold (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Susanne Arnold, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-H&N-11-BMS
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2014-01-23 (Estimated); Last update posted 2023-05-16 (Actual); Status verified 2023-04

CONDITIONS: Squamous Cell Carcinoma
Keywords: head and neck; squamous cell carcinoma; squamous cell; carcinoma; paclitaxel; carboplatin; radiotherapy; induction therapy
MeSH Terms: conditions — Carcinoma, Squamous Cell; Carcinoma | interventions — Radiotherapy; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Induction chemotherapy and radiation (Experimental): Induction chemotherapy with low dose radiation
  Interventions: Radiation: Radiotherapy; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Radiation: Radiotherapy — 80 centigray (cGy) on Day 1 & 2 and 22 & 23 of chemotherapy
Drug: Paclitaxel — 225 mg/m2 intravenously over three hours on Days 1 and 22
  Other Names: Taxol
Drug: Carboplatin — Area under the curve (AUC) of 6 will be given intravenously over 30 minutes on days 1 and 22
  Other Names: Paraplatin, CBDCA

SUMMARY:
This study utilizes two cycles of Paclitaxel and Carboplatin chemotherapies followed by four small doses of radiation, prior to other treatment (surgery or radiation). This study is evaluating if radiation as a chemoenhancer increases the response rate of initial therapy.

DETAILED DESCRIPTION:
Cancers of the head and neck (H&N) comprise 5% of all cancers, with 40,000 new cases diagnosed annually. Surgery followed by irradiation or irradiation alone has been the standard of care for locally advanced Stage III and IV patients. With this approach, fewer than 30% of patients achieve long-term remission, and most recur locoregionally. Neoadjuvant chemotherapy has been administered prior to definitive therapy with response rates ranging from 60-90%; with pathologic complete response (CR) rates documented in 30-70% of clinical responders. However, large randomized trials have shown no improvement in overall survival.

Because induction chemotherapy alone does not appear to improve long-term disease free survival in advanced head and neck cancers, concomitant chemotherapy and radiation has been pursued in patients with locally advanced head and neck cancers. Improved disease-free survival has been demonstrated with a variety of agents. The concept of synergy between radiation and chemotherapy is well established in vitro. Various schedules of radiation and chemotherapy have been utilized including weekly chemotherapy during radiation, chemotherapy given every three weeks during hyperfractionated radiation and alternating chemotherapy and radiation.

One exciting new chemotherapeutic agent, Paclitaxel has been shown to radiosensitize cancer cell lines in vitro. Recent studies have added Carboplatin to Paclitaxel in tandem or concurrently with radiation in hopes of improving response rates. From in-vitro data, it appears that the optimum schedule for the combination of Paclitaxel and radiation is to first induce G2/M arrest with Paclitaxel and follow this with radiation therapy. In a recent study by Chendil, et al, a novel radiation scheme appeared to enhance the response of both p53 wild type and p53 mutant cancer cell lines to chemotherapy. In vitro data with Carboplatin also indicates an additive effect when given prior to irradiation using various cell lines. What has not been evaluated, is whether a neoadjuvant regimen of Paclitaxel and Carboplatin followed by 4 small fractions of radiation can be given safely and effect an improved response rate in patients with bulky T2, Stage III and IV H&N cancer. We propose the use of two cycles of Paclitaxel and Carboplatin followed by four small fractions of radiation, prior to definitive treatment (surgery or radiation). It is hoped that using radiation as a chemoenhancer will increase the response rate to induction therapy in this population of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients greater than 18 years of age.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
3. Patients with pathologically documented bulky T2, III and IV squamous cell cancer of the head and neck (excluding M1 disease), within 2 months of diagnosis. Bulky T2 tumors are defined as those that have a volume of disease greater than 35 cm3 as measured by CT or MRI scan (26).
4. Patients will be medically fit for undergoing chemotherapy. Specifically:

   1. no evidence of active angina pectoris or ventricular arrhythmias; no myocardial infarction within the last six months. (Patients with medically controlled hypertension or congestive heart failure are eligible.)
   2. an absolute neutrophil count of > 1000/uL and platelet count > 100,000/microliter (uL)
   3. serum total bilirubin < 1.5 mg/dL
   4. Creatinine Clearance greater than 50 ml/min

      Using an actual or calculated creatinine clearance using the formula:

      (140 - age) x (wgt in kg)*/(serum creatinine)x(72)*= multiply by 0.85 for females
   5. if a pre-existing grade I neuropathy exists, patients must be willing to risk worsening neuropathy secondary to Paclitaxel. Patients with grade II or greater neuropathy will be excluded from study.
   6. ability to give written, informed consent to participate in the trial.
5. Patients will have measurable disease as determined by MRI or CT scan or evaluable disease determined by panendoscopy to be eligible for enrollment on this study.

Exclusion Criteria:

1. Pregnant females. Males and women of childbearing potential must use effective contraception in order to prevent pregnancy during therapy.
2. Patients with a history of previous or current malignancy at other sites diagnosed within the last 5 years, with the exception of adequately treated carcinoma in-situ of the cervix or basal or squamous cell carcinoma of the skin. Patients with a history of other malignancies, who remain free of recurrence or metastases for greater than five years are eligible.
3. Patients with active infection will not be eligible for this protocol until the infection is treated and the symptoms have clinically resolved.
4. Patients with a history of allergy to drugs utilizing Cremophor in the formulation.
5. Prior induction chemotherapy, prior irradiation or surgery will not be allowed.
6. Patients with metastatic disease will not be eligible for this study.
7. Patients with grade II or greater peripheral neuropathy will be excluded from study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2000-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Arnold, MD, Principal Investigator — University of Kentucky

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of Recruitment: July 2000-May 2002. All patients were recruited from University of Kentucky Markey Cancer Center
Groups:
- Treatment Arm: Induction LDFRT and Chemotherapy: Carboplatin : AUC of 6 will be given intravenously over 30 minutes on days 1 and 22
  Paclitaxel : 225 mg/m^2 intravenously over three hours on Days 1 and 22
  Radiotherapy : 80 cGy on Day 1 & 2 and 22 & 23 of chemotherapy
Period: Overall Study
Arm/Group | Treatment Arm: Induction LDFRT and Chemotherapy
Started | 40
Completed | 39 (1 patient only received 1 cycle and refused further induction, another progressed in neck nodes)
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: Induction LDFRT and Chemotherapy: Carboplatin : AUC of 6 will be given intravenously over 30 minutes on days 1 and 22
  Paclitaxel : 225 mg/m2 intravenously over three hours on Days 1 and 22
  Radiotherapy : 80 cGy on Day 1 & 2 and 22 & 23 of chemotherapy
Arm/Group | Treatment Arm: Induction LDFRT and Chemotherapy
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: Years] | 54 [36 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Response Rate to Induction Chemotherapy Prior to Definitive Therapy (Surgery or Radiation)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: assessed pre-study and once between days 36-57
Measure: Number; unit: participants
Arm/Group | Treatment Arm: Induction LDFRT and Chemotherapy
Number analyzed (Participants) | 39
participants | 32 [0.66 to 0.92]

2. Secondary Outcome: Frequency of Severe (>/= Grade 3) Toxicities
Time Frame: assessed starting on day 1 through study day 58 or until toxicity resolves
Population: Intent to Treat
Measure: Number; unit: adverse events
Arm/Group | Treatment Arm: Induction LDFRT and Chemotherapy
Number analyzed (Participants) | 40
adverse events | 36

3. Secondary Outcome: 5 Year Overall Survival Rates
Time Frame: 5 years post study
Measure: Number; unit: participants
Arm/Group | Treatment Arm: Induction LDFRT and Chemotherapy
Number analyzed (Participants) | 39
participants | 24 (0.0779)

4. Secondary Outcome: 5 Year Disease-specific Survival
Description: Outcome is calculated from the time of enrollment to the time of death due to disease under study or survival to 5 years without death from disease under study, whichever occurs first.The 5-year rates of disease-specific survival were calculated using the Kaplan-Meier method.
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Treatment Arm: Induction LDFRT and Chemotherapy
Number analyzed (Participants) | 39
participants | 26

5. Secondary Outcome: 5 Year Progression Free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Treatment Arm: Induction LDFRT and Chemotherapy
Number analyzed (Participants) | 39
participants | 23

ADVERSE EVENTS:
Arm/Group | Treatment Arm: Induction LDFRT and Chemotherapy
Serious Adverse Events (participants affected / at risk) | 16/40
Other Adverse Events (participants affected / at risk) | 35/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm: Induction LDFRT and Chemotherapy (N=40)
Neutropenia (Infections and infestations) | 15
Infection/Fever (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm: Induction LDFRT and Chemotherapy (N=40)
Neutropenia (Infections and infestations) | 10
Anemia (General disorders) | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Infection/Fever (Infections and infestations) | 12
Arthralgias/myalgias (General disorders) | 21
Nausea (General disorders) | 17
Alopecia (General disorders) | 28
GI (Gastrointestinal disorders) | 4 — GI adverse event includes the following: Diarrhea, constipation, abdominal pain
Mucositis (General disorders) | 5
Neuromotor (Nervous system disorders) | 3
Fatigue (General disorders) | 4
Dysuria (General disorders) | 4
Dermatologic (Skin and subcutaneous tissue disorders) | 3
Pulmonary (General disorders) | 2
Weight Loss (General disorders) | 2

LIMITATIONS AND CAVEATS:
Heterogeneity of post-induction treatment given. While definitive therapy did differ, it was stratified by response to induction therapy, an accepted practice. Conclusions remain exploratory, because of the small sample size and heterogeneity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No